CLINICAL TRIAL: NCT04061226
Title: Relationship Between Normal-weight Central Obesity and Obstructive Sleep Apnea. The Role of Body Fat Distribution in the Prevalence of Obstructive Sleep Apnea.
Brief Title: Relationship Between Normal-weight Central Obesity and Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2014-21
Record Dates: First submitted 2019-08-14; First posted 2019-08-19 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Sleep Disorder; Body Fat Distribution
Keywords: obstructive sleep apnea, normal weight obesity
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Central obesity group: Normal weight central obesity patients (by BMI and WHR).
  Interventions: Device: Overnight polysomnography
- Without central obesity group: Normal weight patients without central obesity (by BMI and WHR).
  Interventions: Device: Overnight polysomnography

INTERVENTIONS:
Device: Overnight polysomnography — Overnight polysomnography will be performed in a sleep laboratory (EEG, EOG, EMG, ECG, respiratory movements of the chest and abdomen, oro-nasal airflow, and O2 saturation will be examined

SUMMARY:
Comparison of the prevalence of obstructive sleep apnea (OSA), measured by polysomnography in normal weight patients with central obesity by body mass index (BMI) and waist hip ratio (WHR), with normal weight patients without central obesity by BMI and WHR.

Evaluation of arterial stiffness and vascular age in normal weight patients with central obesity and in normal weight patients without central obesity.

Determination of the exercise response characteristics in OSA patients.

DETAILED DESCRIPTION:
Body composition (the distribution of adipose tissue) appears to be a risk factor for the prevalence of obstructive form of sleep apnea. The investigators expect a higher prevalence of this serious sleep pathology in normal weight patients with central obesity than in normal weight patient without central obesity. In normal weight patients with central obesity also endothelial dysfunctions, abnormal exercise response to dynamic load and abnormal circadian patterns of blood pressure and heart rate can be expected. There are theoretical assumptions for this hypothesis but relevant studies on sufficiently large samples of patients have not been done. The investigators will also compare the lipid profile in normal weight patients with central obesity with those of normal weight patients without central obesity.

ELIGIBILITY:
Inclusion Criteria central obesity group:

* BMI 18.5 - 24.9 kg/m2 for both men and women
* WHR more than 0.9 for men and 0.85 for women
* no history of myocardial infarction, stroke, atrial fibrillation, previous diagnosis of OSA or its treatment.

Inclusion Criteria without central obesity group:

* BMI 18.5 - 24.9 kg/m2 for men and women
* WHR selected from the lowest tertile of WHR distribution for both men and women

Exclusion Criteria:

* acute infection
* known diagnosis of chronic renal or cardiac failure
* taking drugs that affect sleep (stimulants, hypnotics, antidepressants, antipsychotics, anxiolytics, antihistamines, corticosteroids, theophylline, anti-parkinsonic drugs, anticonvulsants, morphine-type analgetics)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group of patients with normal weight central obesity and group of patients with normal weight without central obesity.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index | Through study completion, an average of 1 year
  Apnea hypopnea index will be measured in both groups

SECONDARY OUTCOMES:
Cardio Ankle Vascular Index (CAVI) | Through study completion, an average of 1 year
  Noninvasive arterial stiffness and vascular age index CAVI will be measured in both groups
Response on ergo-spirometry test | Through study completion, an average of 1 year
  Cardiopulmonary exercise test parameters (oxygen consumption at peak exercise (ml/kg/min) and VE/VCO2 slope) will be measured in both groups.
Ambulatory 24-hour blood pressure measurement (ABPM) | Through study completion, an average of 1 year
  Ambulatory 24-hour blood pressure measurement (ABPM) will be analyzed conventionally and chronobiologically in both broups

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Homolka, M.D.,Ph.D., Principal Investigator — St Anne's University Hospital in Brno
Locations (1):
- St. Anne's University Hospital, Brno, Czechia